CLINICAL TRIAL: NCT06785935
Title: Ultrasound-guided Percutaneous Release of A1 Pulley by a Needle Knife Versus Ultrasound-guided Corticosteroid Injection in the Treatment of Trigger Finger: a Randomized Clinical Trial
Brief Title: Comparison Between 2 Treatment Modalities of Trigger Finger: Ultrasound-guided Percutaneous Release of A1 Pulley by a Needle Knife Versus Ultrasound-guided Corticosteroid Injection in the Treatment of Trigger Finger
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University Hospital (Other)
Responsible Party: Principal Investigator, Nouran Khalid Ibrahim Sallam, Resident of Rheumatology, rehabilitation, and physical medicine department at Mansoura University Hospitals, Mansoura University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS.24.10.2929
Record Dates: First submitted 2025-01-15; First posted 2025-01-21 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2024-12

CONDITIONS: Trigger Finger
MeSH Terms: conditions — Trigger Finger Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients undergoing ultrasonography-guided percutaneous A1 pulley release using a needle knife (Active Comparator)
  Interventions: Device: Needle knife
- Patients undergoing ultrasonography-guided corticosteroid injection under the A1 pulley (Active Comparator)
  Interventions: Drug: Corticosteroid: Betamethasone

INTERVENTIONS:
Device: Needle knife — ultrasonography-guided percutaneous A1 pulley release using a needle knife
  Arms: Patients undergoing ultrasonography-guided percutaneous A1 pulley release using a needle knife
Drug: Corticosteroid: Betamethasone — ultrasonography-guided corticosteroid injection under the A1 pulley
  Arms: Patients undergoing ultrasonography-guided corticosteroid injection under the A1 pulley

SUMMARY:
Trigger finger is a common cause of hand disability and pain in the general population. It is a pathologic condition of the digital pulleys and flexor tendons. Although the pathogenesis is incompletely clear and multifactorial, the most common cause of the trigger finger is the thickened flexor tendon and/or thickened first annular (A1) pulley located at the metacarpophalangeal joint. Currently, ultrasound is considered an effective and valuable tool for assessing the trigger finger, providing static and dynamic evaluations of this condition and a comparison with the adjacent normal digits. Recently, it has been reported that ultrasound-guided percutaneous A1 pulley precise release using a needle knife has received increasing attention in the clinical treatment of trigger fingers and achieved good results. To our knowledge, this is the first clinical study comparing the efficacy and safety of ultrasonic-guided percutaneous A1 pulley release with a needle knife and the ultrasonic-guided steroid injection in treating trigger fingers.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic trigger finger
* Trigger finger at the level of A1 pulley
* Trigger finger of Green's grades II or III

Exclusion Criteria:

* Patients with secondary causes of trigger fingers like diabetes mellitus, rheumatoid arthritis, gout, hypothyroidism, amyloidosis, and sarcoidosis.
* Patients with a previous history of first annular pulley release or injection.
* Patients with trigger fingers of Green's grade I and IV.
* Patients with trigger fingers at any level other than the A1 pulley.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-11-11 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Pain intensity using the visual analog scale (VAS) scoring system | Before the procedure as well as after one week, one month, and three months
Functional ability according to the standard quick disabilities of the arm, shoulder, and hand score (Q DASH) questionnaire | Before the procedure as well as after one week, one month, and three months
Recurrence: The grade of trigger finger according to Green's classiﬁcation | Before the procedure as well as after one week, one month, and three months
Complications such as inflammation, infection, scarring, wound healing problems, and sensory changes | After one week of the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University Hospitals, Al Mansurah, Egypt